CLINICAL TRIAL: NCT06317610
Title: Development and Validation of Growth Prediction Model for Ovarian Cancer Organoids Based on Bright Field Image and Deep Learning
Brief Title: Artificial Intelligence Model for Growth Prediction of Ovarian Cancer Organoids
Status: Recruiting | Type: Observational
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CQGOG0206
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: growth prediction of ovarian cancer organoids in the frame of bright field image by leveraging AI — biopsy or puncture: Patients received biopsy or puncture to obtain tumor tissues or Malignant effusion for organoids establishment

SUMMARY:
The present study aims to collect early bright field image of patient-derived organoids with ovarian cancer. By leveraging artificial intelligence, this study will seek to construct and refine algorithms that able to predict growth of ovarian cancer organoids.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of epithelial ovarian cancer
* Patients received biopsy or puncture to obtain tumor tissues or malignant effusion
* Patients voluntarily participated in the study and signed informed consent.

Exclusion Criteria:

* Non-epithelial ovarian cancer
* No sufficient amount of tumor tissues or malignant effusion for organoids establishment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only women get ovarian cancer
Study Population: Patients with epithelial ovarian cancer received biopsy or puncture to obtain tumor tissues or malignant effusion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
AUC of growth prediction performance using deep learning model | up to 3 years
  AUC =Area under receiver operating characteristic curve
Accuracy of growth prediction using deep learning model | up to 3 years
  Accuracy=( the number of correctly classified samples)/( the number of total samples)

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No